CLINICAL TRIAL: NCT01483508
Title: Contribution of Dietary Cocoa Procyanidins to the Systemic Presence of Flavanols Metabolites in Humans
Brief Title: Absorption and Metabolism of Dietary Cocoa Procyanidins in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 200513038
Record Dates: First submitted 2011-11-28; First posted 2011-12-01 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: flavanols; procyanidins; absorption; cocoa polyphenols; Flavanol and procyanidin absorption in healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Flavanol and procyanidins (Active Comparator)
  Interventions: Other: Flavanol- and procyanidins-containing drink
- Flavanols only (Experimental)
  Interventions: Other: Flavanol-containing drink
- Procyanidins only (Experimental)
  Interventions: Other: Procyanidins-containing drink

INTERVENTIONS:
Other: Flavanol- and procyanidins-containing drink — Single oral intake of a cocoa-based dairy drink containing flavanols [monomer] and procyanidins [dimers to decamers]
  Other Names: Cocoa-based dairy drink
  Arms: Flavanol and procyanidins
Other: Procyanidins-containing drink — Single oral intake of a ocoa-based dairy drink containing procyanidins [dimers to decamers]
  Other Names: Cocoa-based dairy drink
  Arms: Procyanidins only
Other: Flavanol-containing drink — Single oral intake of a cocoa-based dairy drink containing flavanols [monomers]
  Other Names: cocoa-based dairy drink
  Arms: Flavanols only

SUMMARY:
The purpose of this study is to determine whether or not the intake of dietary procyanidins (oligomers of flavanols) contribute to the systemic presence of flavanols in healthy humans.

DETAILED DESCRIPTION:
Flavanols and their oligomeric derivatives, the procyanidins, are plant-derived compounds normally present in the human diet. Accumulating data demonstrate a causal role for flavanols in mediating the cardiovascular benefits associated with the consumption of flavanol-/procyanidin-containing foods. Evidence for a direct, causal role for procyanidins in this context is far less profound. As this is often based on the poor absorption of procyanidins, it has been proposed that procyanidins may indirectly contribute to the systemic presence of bioactive compounds via derivatives generated from the breakdown or catabolism of procyanidins in the gastrointestinal tract. These postulated 'breakdown products' include: i) flavanols, putatively generated by acid hydrolysis in the stomach, and ii) series of phenolic compounds, including 5-(3,4-dihydroxyphenyl)-gamma-valerolactone, that are produced from procyanidin catabolism by the gut microbiome. Verification or rejection of these suppositions could significantly impact the interpretation of epidemiological-/dietary intervention data, and the design of food-content data bases. To address this question, healthy volunteers will consume specially designed cocoa-based dairy drinks containing flavanols and procyanidins (dimers to decamers) either together or individually.

ELIGIBILITY:
Inclusion Criteria:

* A normal blood chemistry and liver function
* Fasting blood cholesterol and triglycerides < 300 mg/dl and < 3.0 mmol/l, respectively
* BMI < 30 kg/m2 will be considered.
* Volunteers must be able to read and speak English fluently, and thus, fully understand the researchers, research protocols, and their rights as a research volunteer.

Exclusion Criteria:

* A history of cardiovascular disease, stroke, uncontrolled hypertension (> 160/90 mm), renal, hepatic, or thyroid disease, GI tract disorders, previous GI surgery, metabolic syndrome, diabetes, taking cholesterol-lowering medication, hormone replacement therapy, antioxidant supplements, on aspirin therapy or taking anticoagulants, or on a medically prescribed diet.
* A history of psychiatric illness or an allergy to peanuts.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Area under the curve described by the concentration of flavanol metabolites in plasma versus time | After consumption at time points 0, 1, 2 and 4 h
  The concentration of flavanol metabolites in plasma is expressed in nmol/L. Flavanol metabolites encompass a series of O-sulfonated, O-glucuronidated and O-methylated flavanol derivatives generated in the gastrointestinal tract and liver after flavanol absorption.
Peak plasma concentration of flavanol metabolites | After consumption at time points 0, 1, 2 and 4 h
  The concentration of flavanol metabolites in plasma is expressed in nmol/L. Flavanol metabolites encompass a series of O-sulfonated, O-glucuronidated and O-methylated flavanol derivatives generated in the gastrointestinal tract and liver after flavanol absorption.

SECONDARY OUTCOMES:
Amount of flavanol metabolites excreted in urine | urine collected up to 24h post-consumption
  The amount of flavanol metabolites excreted in urine is expressed in µmol. Flavanol metabolites encompass a series of O-sulfonated, O-glucuronidated and O-methylated flavanol derivatives generated in the gastrointestinal tract and liver after flavanol absorption.
Amount of 5-(3,4-dihydroxyphenyl)-gamma-valerolactone metabolites in urine | urine collected up to 24 h post-consumption
  The amount of 5-(3,4-dihydroxyphenyl)-gamma-valerolactone metabolites excreted in urine is expressed in µmol. 5-(3,4-dihydroxyphenyl)-gamma-valerolactone metabolites encompass a series of O-sulfonated and O-glucuronidated derivatives generated in the gastrointestinal tract and liver after 5-(3,4-dihydroxyphenyl)-gamma-valerolactone absorption.

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Study Chair — Department of Nutition, University of California Davis; Javier I Ottaviani, PhD, Principal Investigator — Department of Nutrition, University of California Davis
Locations (1):
- Ragle Facility-UC Davis, Davis, California, United States

REFERENCES:
- [Background] Heiss C, Keen CL, Kelm M. Flavanols and cardiovascular disease prevention. Eur Heart J. 2010 Nov;31(21):2583-92. doi: 10.1093/eurheartj/ehq332. Epub 2010 Sep 18. PMID 20852295
- [Background] Manach C, Williamson G, Morand C, Scalbert A, Remesy C. Bioavailability and bioefficacy of polyphenols in humans. I. Review of 97 bioavailability studies. Am J Clin Nutr. 2005 Jan;81(1 Suppl):230S-242S. doi: 10.1093/ajcn/81.1.230S. PMID 15640486
- [Background] Crozier A, Del Rio D, Clifford MN. Bioavailability of dietary flavonoids and phenolic compounds. Mol Aspects Med. 2010 Dec;31(6):446-67. doi: 10.1016/j.mam.2010.09.007. Epub 2010 Sep 18. PMID 20854839
- [Background] Rios LY, Bennett RN, Lazarus SA, Remesy C, Scalbert A, Williamson G. Cocoa procyanidins are stable during gastric transit in humans. Am J Clin Nutr. 2002 Nov;76(5):1106-10. doi: 10.1093/ajcn/76.5.1106. PMID 12399286
- [Background] Holt RR, Lazarus SA, Sullards MC, Zhu QY, Schramm DD, Hammerstone JF, Fraga CG, Schmitz HH, Keen CL. Procyanidin dimer B2 [epicatechin-(4beta-8)-epicatechin] in human plasma after the consumption of a flavanol-rich cocoa. Am J Clin Nutr. 2002 Oct;76(4):798-804. doi: 10.1093/ajcn/76.4.798. PMID 12324293
- [Background] Gonthier MP, Donovan JL, Texier O, Felgines C, Remesy C, Scalbert A. Metabolism of dietary procyanidins in rats. Free Radic Biol Med. 2003 Oct 15;35(8):837-44. doi: 10.1016/s0891-5849(03)00394-0. PMID 14556848
- [Derived] Ottaviani JI, Kwik-Uribe C, Keen CL, Schroeter H. Intake of dietary procyanidins does not contribute to the pool of circulating flavanols in humans. Am J Clin Nutr. 2012 Apr;95(4):851-8. doi: 10.3945/ajcn.111.028340. Epub 2012 Feb 29. PMID 22378733